CLINICAL TRIAL: NCT06404320
Title: Remotely Delivered Physical Activity Program for Treatment-Resistant Depression: A Pilot Randomized Controlled Trial
Brief Title: Physical Activity Program for TRD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-069
Record Dates: First submitted 2024-04-29; First posted 2024-05-08 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Treatment-resistant Depression; Major Depressive Disorder
Keywords: Major Depressive Disorder; Physical Activity; Exercise
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PA program (Experimental): Participants in the PA group will receive a 4-week remotely delivered one-on-one individualized PA program adjunct to TAU.
  Interventions: Behavioral: PA program - MoveU.HappyU
- TAU (No Intervention): Participants in the TAU group will be given a handout with the Canadian 24-hour movement guidelines and be told that they are encouraged to engage in PA.

INTERVENTIONS:
Behavioral: PA program - MoveU.HappyU — Participants will meet with their program trainer once a week virtually for 4 weeks to engage in 30 minutes of behavioral change coaching and 30 minutes of a structured PA program that is tailored to their needs and goals. The intensity of the PA sessions will be self-selected. PA sessions will involve a warmup, a conditioning component consisting of individualized aerobic or resistance exercises, and a cool down/stretch.
  Participants will also be instructed to independently engage in PA (outside of their session with the trainer) for 120 minutes at 50-65% of their maximum work capacity. This can be done by engaging in PA between 3-5 times per week.
  Arms: PA program

SUMMARY:
This is a pilot study examining the delivery of a remotely delivered, one-on-one, individualized physical activity (PA) program in adult participants with treatment-resistant depression (TRD).

DETAILED DESCRIPTION:
More than one-third of patients with major depressive disorder will not respond to at least two antidepressant medication trials, meeting the criteria for TRD. As a result, alternative therapeutic modalities, such as PA, are garnering interest. Numerous studies have reported an association between PA and improvements in mood and mental health. The MoveU.HappyU PA program is an initiative that considers individuals' PA preferences and priorities and works collaboratively to develop individualized PA programs. The program has been found to improve depressive symptoms in a non-clinical sample of university students.

This is a single-site, pilot, randomized controlled clinical trial. The trial will evaluate the feasibility of randomizing adult participants with TRD to a remotely delivered one-on-one individualized PA program (MoveU.HappyU) in addition to treatment as usual (TAU) or TAU. The trial will also assess the acceptability of the PA program and collect data to monitor the efficacy of the PA program for depressive and anxiety symptoms as well as quality of life. This trial includes the use of a digital platform to evaluate the effect of the PA program on passive physiological data that are collected through the use of a wearable device.

Thirty participants will be randomized in a 2:1 allocation to one of two treatment arms: 1) TAU with a 4-week remotely delivered, one-on-one, individualized PA program add-on; 2) TAU without the PA program add-on. Participants in both arms will complete the same clinician-administered scales, self-reported mental health questionnaires, and use a wearable device. After the 4-week interventional period, participants will enter a 6-week observational follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Sedentary adults (engage in less than 60 minutes of moderate-to-vigorous PA per week) between the ages of 18 and 65 years, inclusive, capable of giving informed consent.
2. Participants meeting diagnostic criteria for major depressive disorder without psychotic symptoms according to the Diagnostic and Statistical Manual of Mental Disorders - 5th Ed. and currently experiencing a major depressive episode (MDE) as confirmed by the Mini International Neuropsychiatric Interview (MINI).
3. A Montgomery-Åsberg Depression Rating Scale total score of ≥ 7 at screening (mild-to-severe MDE).
4. Failure of at least two trials of antidepressant therapy of adequate dose and duration during the current episode as established by the Antidepressant Treatment History Form and self-report.
5. Receiving treatments congruent with Canadian Network for Mood and Anxiety Treatments guidelines with no changes to treatments one month before screening (28 days).

Exclusion Criteria:

1. Current symptoms of mania, hypomania, mixed episodes, or psychosis.
2. Have received a diagnosis of alcohol or a substance use disorder within the past 3 months or as confirmed by the MINI. Other secondary psychiatric comorbidities (e.g., anxiety disorders, trauma-related disorders, etc.) will not be excluded.
3. Pregnant females.
4. Acute risk for a cardiovascular event (i.e., cardiovascular event in the past within the past 12 months).
5. Have any medical contraindications to exercise according to the Physical Activity Readiness Questionnaire.
6. Self-reported balance, gait, or locomotion difficulties that would preclude participation in a PA program.
7. Have any other condition that, in the opinion of the investigator(s), would adversely affect the subject's ability to complete the study or its measures.
8. Have exercise-induced asthma.
9. Taking medication that interferes with heart rate response to exercise, such as beta blockers.
10. Do not own a smartphone.
11. Do not have reliable access to the Internet.
12. Have previously received intravenous ketamine treatment in the last 2 months.

Non-English-speaking individuals are excluded because the ability to communicate study information, answer questions accurately and completely about the study, and obtain consent are necessary.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 13 weeks
  Recruitment rate, withdrawal rate, adherence rate, and data completion rate
Acceptability | 13 weeks
  Responses to an exit survey
Acceptability | 13 weeks
  Responses to semi-structured qualitative interviews

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale-17 | 13 weeks
  This is a semi-structured interview that has been well-validated in measuring the presence and severity of depression. This scale will be administered at baseline, at the end of the intervention phase, and at the last follow-up assessment. Scores range from 0 to 52. A decrease in total scores is defined as improvement in depressive symptoms.
Patient Health Questionnaire-9 | 13 weeks
  This scale is a self-rated measure of depressive symptom severity over the past two weeks. This scale will be administered at baseline, at the end of the intervention phase, and at the last follow-up assessment. Scores range from 0 to 27. A decrease in total scores is defined as improvement in depressive symptoms.
General Anxiety Disorder-7 | 13 weeks
  This scale is a self-rated measure of anxiety symptom severity over the past two weeks. This scale will be administered at baseline, at the end of the intervention phase, and at the last follow-up assessment. Scores range from 0 to 21. A decrease in total scores is defined as improvement in anxiety symptoms.
World Health Organization - Five Well-Being Index | 13 weeks
  This scale is a self-rated measure of well-being over the past two weeks. This scale will be modified for weekly administration. The sum of scores from the five items will be multiplied by 4, representing the participant's perceived quality of life as a percentage. Higher scores denote higher quality of life.

OTHER OUTCOMES:
Total duration of sleep; awake, light, rapid eye movement, and deep sleep durations | 13 weeks
  This outcome will be used to assess the effect of the PA program on digital physiological passive data relating to sleep, which will be collected through the use of a wearable device.
Metabolic equivalent minutes | 13 weeks
  This outcome will be used to assess the effect of the PA program on digital physiological passive data relating to activity, which will be collected through the use of a wearable device.
Readiness (interpreted from sleep, activity, resting heart rate, heart rate variability, recovery index, and body temperature scores) | 13 weeks
  This outcome will be used to assess the effect of the PA program on digital physiological passive data relating to readiness, which will be collected through the use of a wearable device.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tassone VK, Quesnel DA, Parkington K, Rueda A, Martin J, Lee GH, Teixeira A, deJonge ML, Lou W, Wiljer D, Mulsant BH, Sabiston CM, Bhat V. Improving adherence to physical activity in treatment-resistant depression: Protocol for a pilot randomized controlled trial of a remotely delivered program. PLoS One. 2025 Sep 2;20(9):e0330848. doi: 10.1371/journal.pone.0330848. eCollection 2025. PMID 40892783